CLINICAL TRIAL: NCT02912507
Title: An Open Label, Split-tattoo Study Comparing the Safety and Efficacy of the 670nm Picosecond Laser Versus the 755 nm Picosecond Laser for Tattoo Removal
Brief Title: Split-tattoo Study Comparing the Safety and Efficacy of 670nm Picosecond Laser Versus 755 nm for Tattoo Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-16-EN15
Record Dates: First submitted 2016-09-16; First posted 2016-09-23 (Estimated); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Tattoo Removal
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational Enlighten Device (Experimental): Tattoo removal treatments with the investigational Cutera enlighten laser
  Interventions: Device: Cutera enlighten laser
- Cynosure PicoSure 755 nm laser (Active Comparator): Tattoo removal treatments with the Cynosure PicoSure 755 nm laser
  Interventions: Device: CynoSure PicoSure 755nm laser

INTERVENTIONS:
Device: Cutera enlighten laser — high-powered, Q-switched 670nm Picosecond laser system indicated for tattoo removal
  Other Names: 670nm Picosecond Laser
  Arms: Investigational Enlighten Device
Device: CynoSure PicoSure 755nm laser — high-powered, Q-switched Alexandrite system that delivers laser energy in the 755 nm wavelength and has received FDA clearance (K133364) for tattoo and benign pigmented lesion removal.
  Arms: Cynosure PicoSure 755 nm laser

SUMMARY:
Study to evaluate safety and efficacy of treatment with the investigational Cutera enlighten laser for tattoo removal as compared to treatment with the Cynosure PicoSure laser

DETAILED DESCRIPTION:
This is an open-label, split-tattoo, single-center prospective, comparison study in up to 20 male or female subjects, age 18 to 65 years, who desire laser removal of a tattoo containing single or multi-color ink. Subjects will receive laser treatments, and will be followed at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male, 18 to 65 years of age (inclusive).
* Fitzpatrick Skin Type I - VI.
* Target tattoo contains single or multi-color ink.
* Subject must be able to read, understand and sign the Informed Consent Form.
* Must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
* Wiling to cover tattoos with a bandage or clothing; and/or have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treated area starting 2 to 4 weeks before the treatment and/or every day for the duration of the study, including the follow-up period.
* Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes.
* Agree to not undergo any other procedure(s) for tattoo removal during the study (as applicable).
* Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study, and no plans to become pregnant for the duration of the study.

Exclusion Criteria:

* Participation in a clinical trial of a drug or another device in the target area during the study.
* Target tattoo contains only black ink.
* History of allergic reaction to pigments following tattooing.
* History of allergy to local anesthetics.
* History of allergy to topical antibiotics.
* History of malignant tumors in the target area.
* Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, scars, large moles.
* Pregnant and/or breastfeeding.
* Having an infection, dermatitis or a rash in the treatment area.
* Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
* Suffering from coagulation disorders or taking prescription anticoagulation medications.
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
* History of vitiligo, eczema, or psoriasis.
* History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
* History of seizure disorders due to light.
* Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
* History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen
* History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer.
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* Systemic use of corticosteroid or isotretinoin within 6 months of study participation.
* Anytime in life, having have used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* Current smoker or history of smoking within 6 months of study participation.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Lezaic, DO, Principal Investigator — Laser Skin Solutions Jacksonville
Locations (1):
- Laser Skin Solutions Jacksonville, Jacksonville Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Halves or single tattoos treated
Groups:
- Single Arm Treatment - Cutera Enlighten Laser: Full tattoo will be treated with the Cutera enlighten laser
- Split Tattoo Treatment - Cutera Enligthen Laser: Tattoo will be split and treated with the Cutera enlighten laser and the Cynosure PicoSure 755 nm laser.
  The investigational treatment will be assigned to either part A (right/top side) or part B (left/lower side) of the tattoo (based on patient's left and right).
- Split Tattoo Treatment - Cynosure PicoSure 755 nm Laser: Tattoo will be split and treated with the Cynosure PicoSure 755 nm laser.
Period: Overall Study
Arm/Group | Single Arm Treatment - Cutera Enlighten Laser | Split Tattoo Treatment - Cutera Enligthen Laser | Split Tattoo Treatment - Cynosure PicoSure 755 nm Laser
Started | 5; 5 Halves or single tattoos treated | 5; 5 Halves or single tattoos treated | 5; 5 Halves or single tattoos treated
Completed | 1; 1 Halves or single tattoos treated | 1; 1 Halves or single tattoos treated | 1; 1 Halves or single tattoos treated
Not Completed | 4; 4 Halves or single tattoos treated | 4; 4 Halves or single tattoos treated | 4; 4 Halves or single tattoos treated

BASELINE CHARACTERISTICS:
Groups:
- Single Arm Treatment: Full tattoo will be treated with the Cutera enlighten laser
- Split Tattoo Treatment: Tattoo will be split and treated with the Cutera enlighten laser and the Cynosure PicoSure 755 nm laser.
- Total: Total of all reporting groups
Arm/Group | Single Arm Treatment | Split Tattoo Treatment | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Degree of Tattoo Clearing as Assessed by the Investigator (Physician's Global Assessment of Improvement)
Description: Degree of tattoo clearing at 6 weeks post-final treatment as assessed by the Investigator (Physician's Global Assessment of Improvement).
  Higher scores indicate better outcomes 4= Very Significant or Complete Clearing 3= Significant Clearing 2= Moderate Clearing
  1= Mild Clearing 0= No Clearing
Time Frame: 6 weeks post-final treatment, an average of 8 months from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Split Tattoo Treatment- Enlighten: Tattoo will be split and treated with the Cutera enlighten laser
- Split Tattoo Treatment- PicoSure: Tattoo will be split and treated with the Cynosure PicoSure 755 nm laser
Arm/Group | Single Arm Treatment | Split Tattoo Treatment- Enlighten | Split Tattoo Treatment- PicoSure
Number analyzed (Participants) | 1 | 1 | 1
score on a scale | 4 (0) | 4 (0) | 4 (0)

ADVERSE EVENTS:
Time Frame: 6 weeks post final treatment, up to 8 months
Groups:
- Split Tattoo Treatment - Cutera Enlighten Laser: Tattoo will be split and treated with the Cutera enlighten laser and the Cynosure PicoSure 755 nm laser.
  The investigational treatment will be assigned to either part A (right/top side) or part B (left/lower side) of the tattoo (based on patient's left and right).
Arm/Group | Single Arm Treatment - Cutera Enlighten Laser | Split Tattoo Treatment - Cutera Enlighten Laser | Split Tattoo Treatment - Cynosure PicoSure 755 nm Laser
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Treatment - Cutera Enlighten Laser (N=5) | Split Tattoo Treatment - Cutera Enlighten Laser (N=5) | Split Tattoo Treatment - Cynosure PicoSure 755 nm Laser (N=5)
Erythema (Skin and subcutaneous tissue disorders) | 5 | 5 | 5
Edema (Skin and subcutaneous tissue disorders) | 4 | 5 | 5
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT02912507/Prot_SAP_000.pdf